CLINICAL TRIAL: NCT06554340
Title: Targeting Vascular Mechanisms of Functional Outcomes Via Home-based Exercise Training Among Persons With Multiple Sclerosis Who Have Hypertension
Brief Title: Vascular Mechanisms, Functional Outcomes, & Exercise Among Persons With Multiple Sclerosis With Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: University of Illinois at Chicago (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tracy Baynard, Professor and Assoc Vice Provost, Grad Edu, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3616
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Hypertension
Keywords: exercise; blood pressure; mobility; cognition
MeSH Terms: conditions — Multiple Sclerosis; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: The proposed study will use a two-arm RCT design to examine the effect of a home-based exercise training program versus an attention control condition on markers of functional recovery, cognition and mobility disability, in persons with MS with hypertension. The primary outcomes will be cognitive performance via the BICAMS battery and mobility disability via the timed 25-foot walk, with secondary effects designed to understand the potential mechanistic role of BP, arterial stiffness, and endothelial function on functional recovery in response to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based aerobic training (Experimental): A 3-month home-based exercise training intervention comprising cycle ergometry as an aerobic mode of training coupled with behavioral coaching. The regimen will be delivered 3-4 days per week.
  Interventions: Behavioral: Home-based aerobic training
- Attention control (No Intervention): The alternative treatment condition comprises a stretching program with minimal exercise and attention control. This program will be delivered using the same frequency and duration as the intervention. The first session will be conducted under the supervision of visiting study personnel as described above. The stretching exercises will follow the manual provided by the National Multiple Sclerosis Society and the investigators will progressively include more exercises and sets over the 3 months, this too has been standardized and manualized for reproducibility. The investigators will provide the same materials and Internet coaching for the attention control group as for the intervention group but focused on stretching and not on increasing aerobic exercise. The investigators will ask that participants not undertake additional exercise during the study duration and this will be documented through an exercise history, the Godin Leisure-Time Exercise Questionnaire.

INTERVENTIONS:
Behavioral: Home-based aerobic training — The aerobic training will focus on large, dynamic movements of the lower extremities using leg cycling ergometry on an upright cycle ergometer installed in the participant's homes and will progress in duration (10-40 minutes) and intensity (50-70% VO2 peak) over the 3-month intervention period. All participants will start exercise at 50% of VO2peak for 10-min as determined by the exercise test, for the first week, to individualize the exercise prescription. Progression will initially target duration with weekly progressions of 5 min to 30 min of exercise, followed by progression of intensity by 5% per week until 70% is attained, based on patient tolerance of the increased work.
  Arms: Home-based aerobic training

SUMMARY:
The goal of this study is to determine if 12 weeks of cycling exercise training at home will improve three parameters: 1) blood pressure, 2) cognition, and 3) walking ability among persons with multiple sclerosis who have high blood pressure, when compared to a group that engages in a 12-week home-based stretching program.

The main questions this study aims to answer are:

1. Can home-based cycling exercise training improve blood pressure by increasing blood vessel dilation in people with multiple sclerosis?
2. Can cycling exercise training improve cognition and walking mobility in people with multiple sclerosis by improving blood pressure?

The investigators will compare home-based cycling training to stretching to see if cycling training improves cognition, walking mobility, blood pressure, and fitness in people with multiple sclerosis.

Participation in this study will take 13-14 weeks, with participants being randomized (like flipping a coin, a 50-50 chance of being in either group) to the home-based cycling training or the stretching group.

All participants will be asked to

* Visit the laboratory two times, one before the beginning of the intervention (home-base training and stretching group) and one at the end of the intervention.
* During visits, participants will complete tests related to cognition, walking mobility, blood pressure and fitness.

DETAILED DESCRIPTION:
Functionally, the disease pathophysiology of multiple sclerosis (MS) brings about a number of consequences, including cognitive dysfunction and mobility disability, which are two of the most prevalent outcomes of MS. Cognitive impairments typically occur in domains of mental processing speed and working memory and is present in 40-70% of patients with MS based on neuropsychological testing. Cognitive impairment compromises quality of life, activities of daily living, employment, and independent living in persons with MS, and co-occurs with decrements in physical abilities. Mobility disability presents as slowed walking speed and reduced walking endurance and presents in nearly 75% of persons with MS population. Cognitive dysfunction and mobility disability might be worsened through the presence of co-morbid conditions that are manageable through life-style behaviors in MS.

Hypertension is the most prevalent cardiovascular comorbidity in MS and is 25% more common in MS than the general population. Yet, there is truly a dearth of research investigating the unique and understudied population of hypertensives with MS. Importantly, hypertension produces vascular changes causing increased blood pressure (BP) pulsatility. The increased pulsatility has been associated with detrimental changes in the brain in the general population and persons with MS. The investigators have shown that BP pulsatility is inversely associated with mobility in people with MS, and that elevated BP is associated with worse cognition in MS. This suggests that mitigating hypertension and decreasing BP pulsatility through lifestyle behaviors may represent important mechanistic pathways for exerting functional adaptations in cognition and mobility for people with MS.

Physical activity and exercise training are effective approaches for improving vascular hemodynamics and BP in the general population of person with hypertension. The investigators have shown that endothelial function and arterial stiffness, which are two important mechanisms related to hypertension, are associated with physical activity in people with MS. The investigators have further shown that exercise training improves endothelial function, mobility, and cognitive function in people with MS. This suggests that exercise training may improve cognition and mobility through vascular outcomes in persons with MS who have hypertension.

The existing studies that improve cardiovascular fitness, cognitive function, and mobility in persons with MS have been center-based, directly supervised, and prescreened participants for the absence of risk factors for cardiovascular disease (CVD). This severely limits the scalability and reach of exercise interventions for managing the functional consequences of MS, and no exercise studies, to date, have targeted persons with MS who are hypertensive, thus, it is unknown if the results will transfer or work better in this group who are higher risk of CVD-related outcomes. Based on our previous randomized controlled trial (RCT) funded by the National Multiple Sclerosis Society (Grant RG4702A), The investigators are the first to successfully demonstrate that a 12-week home-based aerobic exercise intervention, coupled with internet-based monitoring and behavioral coaching, is safe and feasible among persons with MS and yielded improvements in aerobic fitness, vascular function, and mobility. However, our RCT was conducted in volunteers with MS who were prescreened for CVD risk factors (i.e., excluded persons with CVD-related comorbidities), but serves as a precursor for conducting a similar RCT in persons with cardiovascular comorbidities, such as hypertension. The proposed study aims to address this important gap and underrepresented population.

Our long-term goal involves establishing the scientific basis of home-based exercise training as a therapeutic approach for optimizing functional recovery and quality of life in persons with MS. The objective of this application will follow a RCT design and will evaluate if home-based exercise training can elicit improvements in mechanisms of hemodynamic control related to hypertension and yield clinical benefits for cognition and mobility among persons with MS who have hypertension. This would be the first of its kind RCT ever conducted in persons with MS.

Our central hypothesis is that aerobic exercise training will positively impact cognition and mobility disability (two primary outcomes) and that it will also improve cardiovascular-specific mechanisms of hypertension (secondary outcomes). Exercise training improves hypertension, and hypertension is negatively associated with cognition and mobility in older adults and persons with Alzheimer's disease. The investigators believe that a well-designed aerobic exercise training stimulus is likely to improve hypertension-related mechanisms, which will positively impact cognition and mobility disability in persons with MS, thus improving functional recovery. This central hypothesis will be addressed by pursuing two main specific aims and one exploratory specific aim via a 12-week home-based aerobic exercise training program among persons with MS who have hypertension compared with an attention-control program:

1. Specific Aim 1 is to determine if the intervention improves functional outcomes related to cognition, specifically information processing speed, and mobility in hypertensives with MS. Our working hypothesis is that 12 weeks of aerobic exercise training will improve information processing speed (symbol digits modality test (SDMT) and California Verbal Learning Test-II (CVLT-II)) and attenuate mobility disability (e.g., timed 25-foot walk), which are important markers of functional outcomes.
2. Specific Aim 2 will determine if vascular function and BP improve with exercise training compared with control. Our working hypothesis is that 12 weeks of aerobic exercise training will reduce BP and pulsatility, while also improving vascular-specific mechanisms related to hypertension (e.g., endothelial function and arterial stiffness).
3. Specific Aim 3 is exploratory and will determine if the change in BP and vascular function can account for the change in cognition and/or mobility following exercise training. Our exploratory hypothesis is that changes in vascular function and BP will be associated with changes in cognition and walking mobility.

ELIGIBILITY:
Inclusion Criteria:

* Persons with confirmed multiple sclerosis diagnosis with Expanded Disability Status Scale scores of 4-6.5, characteristic of 2nd stage of multiple sclerosis;
* Hypertension defined as elevated, or Stage 1 or 2, as per the 2017 American Heart Association guidelines (brachial systolic blood pressure > 120 mmHg or brachial diastolic blood pressure > 80 mmHg)
* Persons who are physically inactive (less than 60 min/wk of physical activity);
* Persons with body mass index < 40 kg/m2;
* Persons who are not confined to a wheel chair;
* Multiple sclerosis relapse in the past 30 days;
* People with stable pharmacotherapy.

Exclusion Criteria:

* People with additional cardiovascular comorbidities;
* People with type 1 diabetes mellitus;
* Physician disapproval to participating in the study;
* Space constraints to fit a cycle ergometer at the home of prospective participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Information processing speed | Baseline, pre-intervention/BICAMS; Within 5 days after completion of the training intervention/BICAMS
  The Brief International Cognitive Assessment (BICAMS) battery tests, including the Symbol Digit Modalities Test (SDMT) and California Verbal Learning Test-II (CVLT-II)
Timed 25-Foot Walk | Baseline, pre-intervention/25-Foot Walk; Within 5 days after completion of training intervention/ 25-Foot Walk
  Measurement of mobility disability

SECONDARY OUTCOMES:
Blood pressure | Baseline, pre-intervention/oscillometry, applanation tonometry; Within 5 days after completion of training intervention/oscillometry, applanation tonometry
  24h Blood pressure and central systolic blood pressure
Flow-mediated dilation | Baseline, pre-intervention/ultrasonography; Within 5 days after completion of training intervention/ultrasonography
  Non-invasive measurement of endothelium-dependent vasodilation and macrovascular function
Forearm blood flow | Baseline, pre-intervention/ strain-gauge plethysmography; Within 5 days after completion of training intervention/strain-gauge plethysmography
  Non-invasive measurement of microvascular function
Cardiorespiratory fitness | Baseline, pre-intervention/indirect calorimetry; Within 5 days after completion of training intervention/indirect calorimetry
  Maximal oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fernhall, PhD, Principal Investigator — University of Massachusetts, Boston; Tracy Baynard, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- UMass Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No